CLINICAL TRIAL: NCT05432648
Title: Clinical Tolerance and Microbiome Changes Following Fiber Food Introduction in Short Bowel Syndrome
Brief Title: Fiber Food Introduction in Pediatric Short Bowel Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-019185
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Short Gut Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Bowel Syndrome Arm (Experimental): Patients with SBS will be initiated on green bean purees added to enteral formula recipes, based on kilocalories of enteral formula over 3 weeks. During week 1 subjects will prepare and add 50 mL green bean puree per 1000kcal of enteral feed (5%) to their formula mixture, increasing to 100ml (10%) and 150ml (15%) during weeks 2 and 3, respectively.
  Interventions: Dietary Supplement: Green bean puree
- Control Arm - (Active Comparator): Patients without SBS will be initiated on green bean purees added to enteral formula recipes, based on kilocalories of enteral formula over 3 weeks. During week 1 subjects will prepare and add 50 mL green bean puree per 1000kcal of enteral feed (5%) to their formula mixture, increasing to 100ml (10%) and 150ml (15%) during weeks 2 and 3, respectively.
  Interventions: Dietary Supplement: Green bean puree

INTERVENTIONS:
Dietary Supplement: Green bean puree — Green bean contains both soluble and insoluble fiber, which may have different extent of influence on the gut microbiome. Using a real food rather than a purified fiber such as pectin is more practical and more acceptable to families.

SUMMARY:
Short bowel syndrome (SBS) is a rare but challenging condition in which patients have insufficient bowel length to meet fluid, electrolyte, and nutrient requirements without parenteral support.

The purpose of this study is to determine how well dietary fiber is tolerated in patients with short bowel syndrome compared to patients without short bowel syndrome based on assessment of gastrointestinal symptoms, and corresponding changes in microbiome composition and metabolomics.

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is a rare but challenging condition in which patients have insufficient bowel length to meet fluid, electrolyte, and nutrient requirements without parenteral support. The goal of SBS treatment is to achieve enteral autonomy using strategies that optimize intestinal absorption while minimizing unpleasant gastrointestinal (GI) side effects. One strategy that has emerged is the addition of soluble fiber to enteral formula, and this strategy has gained popularity in clinical practice as fiber-rich formulas comprised of blenderized whole foods have become commercially available. However, the investigators' preliminary observations suggest that patients with SBS have variable tolerance and growth outcomes on these blenderized feeds. To date, there are no clinical studies documenting the effects of dietary fiber in SBS patients and guidance in enteral nutrition advancement is lacking in this medically complex population. The current study aims to explore the tolerance of controlled fiber addition to enteral formula based on assessment of GI symptoms, and corresponding changes in microbiome composition, and metabolomics in pediatric patients with SBS versus non-SBS controls. The investigators will use a practical approach with fiber introduction and slowly advance to goal fiber intake to understand the factors leading to continuation. Stool, urine, and plasma samples collected pre- and post- intervention will help identify biomarkers that would predict successful fiber tolerance and optimize selection of patients for fiber introduction. While there is no intent to treat, mitigate, prevent, diagnose or cure the symptoms of SBS, the study may help shed light on the underlying mechanism for intolerance to dietary fiber.

ELIGIBILITY:
Inclusion Criteria:

* Actively follows at the Children's Hospital of Philadelphia (CHOP) outpatient clinics
* SBS arm specific: History of SBS diagnosis. History of short bowel syndrome based on surgical/imaging records. Small bowel is in continuity with some portion of colon
* Control arm specific: No history of intestinal pathologies
* No or negligible amount (few bites of fiber-containing foods okay) of fiber in tube feeds or by mouth at baseline
* Less than 20% calories from oral food not containing fiber while the other 80% may be by enteral and/or parenteral feedings
* At least 20% calories from fiber-free formula taken orally or via tube
* Antibiotic use is allowed, however, should be on a stable regimen of antibiotics starting from 2 weeks prior to intervention until end of study or end of week 3 whichever is sooner. Instances of antibiotic use for brief courses (7-10 days) as long as sample collection is scheduled to be at least a week from the end date of antibiotics.
* Previous history of fiber introduction failure is acceptable as long as clinically stable at the time of recruitment
* Fiber supplementation is appropriate per primary physician
* If subject is unable to provide full set of samples, they will still be enrolled

Exclusion Criteria:

* SBS Arm specific: No diagnosis of SBS.
* Control Arm specific: has baseline intestinal diseases
* Small bowel and colon not in continuity (Ex: presence of ileostomy or jejunostomy)
* >5% changes in percentage of calories from oral nutrition (PO), enteral nutrition (EN) and/or parenteral nutrition (PN) during the intervention
* Addition/discontinuation/significant alteration to antibiotics regimen during study period
* Primary physician does not think fiber supplementation is appropriate clinically

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-08 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Symptoms | 3 weeks-6 months
  To assess the rate of continuation and symptoms/signs leading to discontinuation of fiber addition in SBS vs controls

SECONDARY OUTCOMES:
Microbiome/Metabolome Changes | 3 weeks-6 months
  To correlate changes in clinical status on fiber to microbiome/metabolome changes in SBS vs controls

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Albenberg, DO, Principal Investigator — Children's Hospital of Philadelphia; Christina Bales, MD, Principal Investigator — Children's Hospital of Philadelphia; Wenjing Zong, MD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States